CLINICAL TRIAL: NCT01768975
Title: Randomized, Double-Blind, Vehicle-Controlled, Efficacy and Safety Clinical Trial of Topically Applied OLT1177 Gel in Subjects With Moderate to Severe Pain Associated With Osteoarthritis of the Knee Following Cessation of Pain Therapy
Brief Title: Phase 2 Efficacy Trial of OLT1177 Gel in Subjects With Moderate to Severe Pain Associated With OA of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Olatec Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OLT1177-02
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-09

CONDITIONS: Osteoarthritis of the Knee
Keywords: Knee; Osteoarthritis; OA; Knee pain; Moderate pain; Severe pain; Inflammation; Safety; Efficacy; Randomized; Topical; Gel; Olatec; OLT1177; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases; Arthritis; Therapeutic; Analgesic
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain; Inflammation; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases; Arthritis | interventions — dapansutrile

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OLT1177 Gel (Experimental): 4 mL per dose, applied 3 times per day on Days 1 - 13 with only one dose administered on Day 14, assuming TID on Day 1
  Interventions: Drug: OLT1177 Gel
- Placebo gel (Placebo Comparator): Identical dose and dosing regimen as the Investigational Drug (OLT1177 Gel)
  Interventions: Other: Placebo gel

INTERVENTIONS:
Drug: OLT1177 Gel — 4 mL per dose, applied 3 times per day on Days 1 - 13 with only one dose administered on Day 14, assuming TID on Day 1
  Other Names: OLT1177
  Arms: OLT1177 Gel
Other: Placebo gel — Identical dose and dosing regimen as the Investigational Drug (OLT1177 Gel)
  Arms: Placebo gel

SUMMARY:
The purpose of this trial is to investigate the efficacy and safety of OLT1177 Gel in subjects with moderate to severe pain associated with osteoarthritis of the knee following cessation of pain therapy.

DETAILED DESCRIPTION:
This is a randomized, double-blind, vehicle-controlled, repeat-dose, multi-center Phase 2 efficacy and safety clinical trial of subjects with moderate to severe pain associated with osteoarthritis of the knee. Eighty-four subjects, randomized in a 2:1 ratio (OLT1177 Gel to vehicle control) will receive up to 40 doses of the Investigational Drug (56 subjects OLT1177 Gel and 28 subjects vehicle control) over 14 consecutive days given 3 times per day (4 mL per dose, TID on Days 1 - 13 with only one dose administered on Day 14, assuming TID on Day 1) and will have safety data collected through Day 28. Subjects with moderate to severe pain associated with osteoarthritis of the knee will be evaluated twice for eligibility: 1) at the Screening visit; and 2) at the Baseline (Day 0) visit, after a 7-day washout period of all pain medications except for trial provided Rescue Medication (500 mg/dose of acetaminophen) for those that experience unacceptable pain during the washout and 14-day treatment period.

Subjects will be encouraged not to take any pain medication during the 7-day washout period; however, for the first 5 days they are allowed to take only Rescue Medication. No pain medication, including Rescue Medication, is allowed during the 2-day pain intensity assessment period or within 48 hours of the Baseline (Day 0), Day 7 and Day 14 visits.

Subjects will be asked to record and report their level of pain at different time points throughout the 14-day trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 35 to 80
* Subjects of childbearing potential and their partners must use effective contraception
* OA based on the ACR criteria
* OA of the knee ≥ 6 months prior to Screening
* OA knee pain which required NSAID or other therapy for ≥ 15 days
* Pain on Movement in the contralateral knee be ≤ 20 mm
* Radiographic evidence of OA by Kellgren-Lawrence score of 2 or 3 taken 6 months prior to Screening
* Moderate to severe OA pain defined as POM score between 50 mm and 90 mm
* Baseline WOMAC pain subscale score ≥ 9
* No change in physical activity and/or therapy for the past 3 months
* Provide written informed consent and comply with the trial

Exclusion Criteria:

* Use of Rescue Medication or any other pain medication 48 hours prior to Baseline visit
* Inflammatory skin condition over the target knee
* Extreme pain in the target knee characterized by POM score of > 90 mm
* Mild pain in the target knee, characterized by POM score of < 50 mm
* > 30 mm POM score variability in Days -2 to -1 from Baseline visit
* Baseline POM score of > 20 mm for the contralateral knee or any other significant joint or general pain at Baseline visit
* Excessive effusion in the target knee
* Heat and/or redness in comparison to the contralateral knee
* Knock-kneed or bow-legged defined by valgus or varus deformity of ≥ 15 degrees
* Acute or chronic injury other than OA
* Radiographic evidence of OA by Kellgren-Lawrence score of 0, 1 or 4
* Open surgery of the target knee within the last year
* Arthroscopic surgery of the target knee within the last 6 months
* Surgery of the target knee requiring insertion of a medical device or surgical hardware
* Use of prohibited concomitant medications/therapies during the 7-day washout period or planned use during the 14-day treatment period including:

  1. Prescription medications to treat pain, OTC and natural supplements
  2. Muscle relaxants unless on a stable dose ≥ 30 days prior to Screening
  3. Nutraceuticals unless on a stable dose ≥ 3 months prior to Screening
  4. Sedative hypnotics unless on a stable dose ≥ 30 days prior to Screening
  5. Devices or therapeutic treatments for knee pain or ambulation
  6. Systemic corticosteroids
  7. Other Investigational Drugs
  8. Chemotherapeutic drugs
  9. Immunotherapy
  10. Topical products applied to the target knee
  11. Cyclosporine (except ophthalmic), lithium, methotrexate
  12. Anti-depressants or medications acting on the central nervous system, unless on a stable dose for depression ≥ 3 months prior to Screening
  13. Narcotics or previous history of chronic narcotic use
  14. Rescue Medication within 48 hours of Baseline, Day 7 or Day 14 visits
* Intraarticular steroids in the target knee within the previous 3 months or in any other joint within the previous 30 days
* Intraarticular hyaluronate within the previous 6 months or in any other joint within the previous 30 days
* Systemic corticosteroids within the prior month
* Documented history of inflammatory joint disease
* BMI over 35
* Uncontrolled psychiatric conditions
* Cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological or neurological disease or prior surgery
* Uncontrolled hypertension
* Diabetes with an HbA1c level > 8
* Known positive for HIV, Hepatitis B surface antigen (HBsAg) or antibodies to Hepatitis C Virus (HCV)
* Cancer within the past 5 years, except for treated basal cell or squamous cell carcinoma of the skin
* Any other medical conditions, diseases or prior surgeries
* Interventional and/or surgical procedure during the 28 days following randomization
* Change in level of physical activity during the 28 days following randomization
* Active infection or fever ≥ 38°C within 3 days of Baseline visit
* Known sensitivity to Investigational Drug
* Women planning to become pregnant during the 28-day trial
* Participation in any Investigational Drug or device trial within 30-day prior to Baseline visit

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in WOMAC knee pain subscale (scale 0 - 20) | 14 days
  The mean group change for OLT1177 Gel and vehicle control from Baseline (Day 0) to Day 14 in WOMAC knee pain subscale (Scale 0-20), which is determined by the subjects responses to five questions (S1-S5) using a 5-point Likert scale (i.e., 'none'=0; 'mild'=1, 'moderate'=2; 'severe'=3; 'extreme'=4)

SECONDARY OUTCOMES:
Change in Current Knee Pain (100-mm VAS) | 50 minutes post dose (± 10 minutes)
  The mean group change in Current Knee Pain (100-mm VAS) for OLT1177 Gel and vehicle control from Baseline (Day 0) pre-dose to Day 1, 50-minutes post-dose (± 10 minutes) calculated in millimeters and percentage, as recorded by the subjects during the Baseline (Day 0) visit after the first application of the Investigational Drug
Mean group rating of Relative Knee Pain (5-point scale) | 50 minutes post dose (± 10 minutes)
  The mean group rating of Relative Knee Pain (5-point scale) for OLT1177 Gel and vehicle control at Day 1, 50-minutes post-dose (± 10 minutes) as recorded by the subjects during the Baseline (Day 0) visit after the first application of the Investigational Drug
Change in WOMAC knee pain subscale | 7 days
  The mean group change for OLT1177 Gel and vehicle control from Baseline (Day 0) to Day 7 in WOMAC knee pain subscale (Scale 0-20), which is determined by the subjects responses to five questions during the Day 7 site visit
Change in Pain on Movement (100-mm VAS) | 7 days
  The mean group change in Pain on Movement (100-mm VAS) for OLT1177 Gel and vehicle control from Baseline (Day 0) to Day 7, calculated in millimeters and percentage, as recorded by the subjects while at home
Change in Pain on Movement (100-mm VAS) | 14 days
  The mean group change in Pain on Movement (100-mm VAS) for OLT1177 Gel and vehicle control from Baseline (Day 0) to Day 14, calculated in millimeters and percentage, as recorded by the subjects while at home
Change in Global Rating of Disease | 14 days
  The mean group change in Global Rating of Disease for OLT1177 Gel and vehicle control from Baseline (Day 0) to Day 14 measured on a 5-point Likert scale, with numerical values to be assigned as follows: 0 = poor, 1 = fair, 2 = good, 3 = very good and 4 = excellent, as recorded by the subjects at the Day 14 site visit
Change in Global Evaluation of Treatment | 14 days
  The mean group rating of Global Evaluation of Treatment for OLT1177 Gel and vehicle control at Day 14 measured on a 5-point Likert scale, with numerical values to be assigned as follows: 0 = poor, 1 = fair, 2 = good, 3 = very good and 4 = excellent, as recorded by the subjects at the Day 14 site visit
Change in WOMAC Stiffness subscale (Scale 0-8) | 7 days
  The mean group change for OLT1177 Gel and vehicle control from Baseline (Day 0) to Day 7 in the WOMAC Stiffness subscale (Scale 0-8) and in the WOMAC Physical function subscale (Scale 0-68), which is determined by subjects responses to questions at the Day 7 site visit
Change in WOMAC Stiffness subscale (Scale 0-8) | 14 days
  The mean group change for OLT1177 Gel and vehicle control from Baseline (Day 0) to Day 14 in the WOMAC Stiffness subscale (Scale 0-8) and in the WOMAC Physical function subscale (Scale 0-68), which is determined by subjects responses to questions at the Day 14 site visit
Change in the use of Rescue Medication | 14 days
  The mean group change for OLT1177 Gel and vehicle control in the proportion of subjects who required the use of Rescue Medication
Change in the time to use of Rescue Medication | 14 days
  The mean group time to use of Rescue Medication for OLT1177 Gel and vehicle control after the first dose of Investigational Drug
Proportion of subjects experiencing an improvement in WOMAC knee pain subscale | 14 days
  The proportion of subjects who experience an improvement in WOMAC knee pain subscale (Scale 0-20, transformed to a 0 to 100 scale) from Baseline (Day 0) to Day 14 equal to or greater than the minimum clinically important improvement (MCII) threshold of 15-mm
Proportion of subjects experiencing an improvement in WOMAC knee pain subscale | 14 days
  The proportion of subjects who experience an improvement in WOMAC knee pain subscale (Scale 0-20, transformed to a 0 to 100 scale) from Baseline (Day 0) to Day 14 equal to or greater than the minimum clinically important improvement (MCII) threshold of 20%
Proportion of subjects whose WOMAC knee pain subscale is less than the PASS | 14 days
  The proportion of subjects whose WOMAC knee pain subscale (Scale 0-20, transformed to a 0 to 100 scale) at Day 14 is less than the patient acceptable symptom state (PASS) of 40
Proportion of subjects experiencing an improvement in Pain on Movement | 14 days
  The proportion of subjects who experience an improvement in Pain on Movement (100-mm VAS) from Baseline (Day 0) to Day 14 equal to or greater than the minimum clinically important improvement (MCII) threshold of 15-mm
Proportion of subjects experiencing an improvement in Pain on Movement | 14 days
  The proportion of subjects who experience an improvement in Pain on Movement (100-mm VAS) from Baseline (Day 0) to Day 14 equal to or greater than the minimum clinically important improvement (MCII) threshold of 20%
Proportion of subjects whose POM is less than the PASS | 14 days
  The proportion of subjects whose Pain on Movement (100-mm VAS) at Day 14 is less than the patient acceptable symptom state (PASS) of 40-mm

CONTACTS AND LOCATIONS:
Overall Officials: Jaime A. Pachon, MD, Principal Investigator — Miami Research Associates; Bruce G. Rankin, D.O., C.P.I, Principal Investigator — Avail Clinical Research; Treva W. Tyson, MD, Principal Investigator — Wake Research Associates
Locations (3):
- United States (3):
  - Avail Clinical Research, DeLand, Florida
  - Miami Research Associates, South Miami, Florida
  - Wake Research Associates, Raleigh, North Carolina